CLINICAL TRIAL: NCT01989156
Title: A Randomized, Controlled, Open-label, 3-arm Parallel Group, Multi-center Study to Demonstrate Reductions in Exposure to Selected Smoke Constituents in Apparently Healthy Smokers Switching to the Tobacco Heating System 2.2 Menthol (THS 2.2 Menthol) or Observing Smoking Abstinence, Compared to Continuing to Use Menthol Conventional Cigarettes, for 5 Days in Confinement and Prolonged by 86 Days in an Ambulatory Setting
Brief Title: Reduced Exposure Study Using THS 2.2 Menthol With 5 Days in a Confinement Setting Followed by 86 Days in an Ambulatory Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZRHM-REXA-08-US; ZRHM-REXA-08-US (Other: Philip Morris Products S.A.)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Smoking
Keywords: Smoking; Candidate modified risk tobacco product; Menthol conventional cigarettes; Reduced exposure; HPHCs; Ambulatory
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- THS 2.2 Menthol (mTHS 2.2) (Experimental): Ad libitum use of THS 2.2 Menthol for 5 Days in a Confinement Setting and 86 Days in an Ambulatory Setting
  Interventions: Other: THS 2.2 Menthol (mTHS 2.2)
- Menthol Conventional Cigarette (mCC) (Active Comparator): Ad libitum use of subject's own preferred brand of mCC for 5 Days in a Confinement Setting and 86 Days in an Ambulatory Setting
  Interventions: Other: Menthol Conventional Cigarette (mCC)
- Smoking abstinence (SA) (Sham Comparator): Abstinence from smoking for 5 Days in a Confinement Setting and 86 Days in an Ambulatory Setting
  Interventions: Other: Smoking Abstinence (SA)

INTERVENTIONS:
Other: THS 2.2 Menthol (mTHS 2.2) — THS 2.2 Menthol ad libitum for 5 days in confinement prolonged by 86 days in an ambulatory setting
  Arms: THS 2.2 Menthol (mTHS 2.2)
Other: Menthol Conventional Cigarette (mCC) — Subject's own preferred brand of mCC ad libitum for 5 days in confinement prolonged by 86 days in an ambulatory setting
  Arms: Menthol Conventional Cigarette (mCC)
Other: Smoking Abstinence (SA) — SA for 5 days in confinement prolonged by 86 days in an ambulatory setting
  Arms: Smoking abstinence (SA)

SUMMARY:
Evaluate if the ad libitum use of the THS 2.2 Menthol (mTHS), a candidate Modified Risk Tobacco Product, for 5 days in confinement, and after 86 days in an ambulatory setting, by apparently adult healthy smokers results in a reduction in the levels of biomarkers of exposure (BoExp) to selected harmful and potentially harmful constituents (HPHCs).

DETAILED DESCRIPTION:
The main goal of the study is to evaluate if the ad libitum use of the THS 2.2 Menthol (mTHS) for 5 days in confinement, and after 86 days in an ambulatory setting, by apparently adult healthy smokers results in a reduction in the levels of biomarkers of exposure (BoExp) to selected harmful and potentially harmful constituents (HPHCs) compared to smokers continuing smoking their own preferred brand of menthol conventional cigarette (mCC) and smoking abstinence (SA). Smokers who remained abstinent from SA were used as a benchmark to provide context to the exposure reduction.

ELIGIBILITY:
Inclusion Criteria:

* Smoking, apparently healthy subject as judged by the Investigator.
* Subject smokes at least 10 commercially available mCCs per day (no brand restrictions) for the last 4 weeks, based on self-reporting.
* Subject has smoked for at least the last 3 consecutive years.
* Subject does not plan to quit smoking within the next 6 months.

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
* The subject has received medication within 14 days or within 5 half-lives of the medication (whichever is longer), which has an impact on CYP1A2 or CYP2A6 activity.
* For women: Subject is pregnant or is breast feeding.
* For women: Subject does not agree to use an acceptable method of effective contraception.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Lewis, MD, Principal Investigator — Covance Dallas; Frank Farmer, MD, Principal Investigator — Covance Daytona Beach; Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.
Locations (2):
- United States (2):
  - Covance Daytona Beach, 1900 Mason Ave., Suite 140, Daytona Beach, Florida
  - Covance Dallas, 1341 W. Mockingbird Ln., Ste 400E, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haziza C, de La Bourdonnaye G, Donelli A, Skiada D, Poux V, Weitkunat R, Baker G, Picavet P, Ludicke F. Favorable Changes in Biomarkers of Potential Harm to Reduce the Adverse Health Effects of Smoking in Smokers Switching to the Menthol Tobacco Heating System 2.2 for 3 Months (Part 2). Nicotine Tob Res. 2020 Apr 17;22(4):549-559. doi: 10.1093/ntr/ntz084. PMID 31125079
- [Derived] Haziza C, de La Bourdonnaye G, Donelli A, Poux V, Skiada D, Weitkunat R, Baker G, Picavet P, Ludicke F. Reduction in Exposure to Selected Harmful and Potentially Harmful Constituents Approaching Those Observed Upon Smoking Abstinence in Smokers Switching to the Menthol Tobacco Heating System 2.2 for 3 Months (Part 1). Nicotine Tob Res. 2020 Apr 17;22(4):539-548. doi: 10.1093/ntr/ntz013. PMID 30722062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (first subject screened): 17 December 2013
  At admission (Day -2), all the subjects performed a product trial of THS 2.2 Menthol. During the baseline period, they continued to smoke their single preferred brand of mCC. Then, on Day 0, they were randomized to one of the 3 study arms (mTHS 2.2, mCC or SA) in a 2:1:1 ratio.
Pre-assignment Details: Enrolled and randomized population = 160 subjects
  * 80 subjects in mTHS 2.2
  * 41 subjects in mCC
  * 39 subjects in SA
  Number of subjects exposed to the product test = 165
  * Number of subjects enrolled but NOT randomized = 4
  * Number of subjects failed screening = 1
Period: Confinement Period (Population at Day 5)
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Started | 80 | 41 | 39
Completed | 80 | 40 | 34
Not Completed | 0 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 3
Not completed — Patient Anxiety | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Period: End of Study (Population at Day 90)
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Started | 80 | 40 | 34
Completed | 73 | 35 | 31
Not Completed | 7 | 5 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Lost to Follow-up | 3 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Moved out of state | 1 | 0 | 0
Not completed — Employment Conflict | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study population = all randomized subjects who had at least one post randomization product use experience and at least one valid biomarker of exposure measurement.
  160 randomized subjects: 80 in mTHS 2.2, 41 in mCC and 39 in SA arms
Groups:
- Total: Total of all reporting groups
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA) | Total
Number analyzed (Participants) | 80 | 41 | 39 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (11.72) | 33.7 (10.17) | 38.8 (11.42) | 37.7 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 17 | 15 | 64
  Male | 48 | 24 | 24 | 96
Daily mCC consumption at screening [Number; unit: participants]
  10 to 19 cig/day | 43 | 21 | 18 | 82
  > 19 cig/day | 36 | 20 | 21 | 77

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Monohydroxybutenylmercapturic Acid (MHBMA)
Description: Concentrations measured in urine, adjusted for creatinine, at Day 5 for the smokers of all arms (mTHS, mCC and SA). Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 5 days
Population: The analysis was performed on the Per Protocol set (PP) which included all randomized subjects who had no major protocol deviation impacting the evaluability during the confinement period.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 65 | 30 | 21
pg/mg creat | 110.96 [93.49 to 131.68] | 882.25 [687.25 to 1132.57] | 94.97 [70.67 to 127.61]
Statistical Analysis 1: Comparison: THS 2.2 Menthol (mTHS 2.2) vs Menthol Conventional Cigarette (mCC); The hypothesis to be tested is that the geometric mean level on Day 5 of the biomarker of exposure for mTHS 2.2 is lower relative to mCC. Analysis of the biomarkers of exposure (BoExp) was conducted on the natural log scale in order to test the following hypothesis (one sided test with 2.5% type I error probability): * Null hypothesis (H0): m1≥m2 * Alternative hypothesis (H1): m1<m2 Where m1 and m2 are the geometric means of the BoExp levels on Day 5 for mTHS 2.2 and mCC respectively; Test type: Superiority or Other; p < 0.001, ANCOVA — The primary endpoints were tested using a multiple testing procedure to preserve the overall alpha level by simultaneously testing the endpoints using a closed procedure with each test performed at an alpha level of 2.5% one sided; ANCOVA model on MHBMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 12.58, 95% CI 2-sided [9.27 to 17.05] — Geometric LS Mean Ratio mTHS 2.2:mCC

2. Primary Outcome: Concentration of 3-hydroxypropylmercapturic Acid (3-HPMA)
Description: as for outcome 1
Time Frame: 5 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mg creat
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 67 | 30 | 21
ng/mg creat | 278.13 [254.95 to 303.43] | 607.68 [534.34 to 691.09] | 152.05 [130.47 to 177.19]
Statistical Analysis 1: Comparison: THS 2.2 Menthol (mTHS 2.2) vs Menthol Conventional Cigarette (mCC); The hypothesis to be tested is that the geometric mean level on Day 5 of the biomarker of exposure for mTHS 2.2 is lower relative to mCC. Analysis of the BoExp was conducted on the natural log scale in order to test the following hypothesis (one sided test with 2.5% type I error probability): * Null hypothesis (H0): m1≥m2 * Alternative hypothesis (H1): m1<m2 Where m1 and m2 are the geometric means of the BoExp levels on Day 5 for mTHS 2.2 and mCC respectively; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on 3-HPMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 45.77, 95% CI 2-sided [39.22 to 53.41] — Geometric LS mean ratio mTHS 2.2:mCC

3. Primary Outcome: Concentration of S-phenylmercapturic Acid (S-PMA)
Description: as for outcome 1
Time Frame: 5 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 65 | 30 | 21
pg/mg creat | 134.11 [114.63 to 156.90] | 1065.91 [848.45 to 1339.09] | 131.05 [99.78 to 172.13]
Statistical Analysis 1: Comparison: THS 2.2 Menthol (mTHS 2.2) vs Menthol Conventional Cigarette (mCC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on S-PMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 12.58, 95% CI 2-sided [9.54 to 16.58] — Geometric LS mean ratio mTHS 2.2:mCC

4. Primary Outcome: Levels of Total 4-(Methylnitrosamino)-1-(3- Pyridyl)-1-butanol (Total NNAL)
Description: Concentrations measured in urine, adjusted for creatinine, at Day 90 for the smokers of all arms (mTHS, mCC and SA). Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 90 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 43 | 29 | 9
pg/mg creat | 41.05 [31.28 to 53.86] | 155.45 [112.46 to 214.88] | 54.03 [30 to 97.28]
Statistical Analysis 1: Comparison: THS 2.2 Menthol (mTHS 2.2) vs Menthol Conventional Cigarette (mCC); The hypothesis to be tested is that the geometric mean level on Day 90 of the biomarker of exposure for mTHS 2.2 is lower relative to mCC. Analysis of the BoExp was conducted on the natural log scale in order to test the following hypothesis (one sided test with 2.5% type I error probability): * Null hypothesis (H0): m1≥m2 * Alternative hypothesis (H1): m1<m2 Where m1 and m2 are the geometric means of the BoExp levels on Day 90 for mTHS 2.2 and mCC respectively; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on Total NNAL levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 26.41, 95% CI 2-sided [17.31 to 40.26] — Geometric LS mean ratio mTHS 2.2:mCC

5. Primary Outcome: Levels of Carboxyhemoglobin (COHb)
Description: Carboxyhemoglobin (COHb) is assayed from whole blood. Expressed as % of saturation of hemoglobin. Blood measurements performed in the evening of Day 5, for the smokers of all arms (mTHS, mCC and SA). Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 5 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: % of saturation of hemoglobin
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 74 | 34 | 23
% of saturation of hemoglobin | 2.33 [2.19 to 2.48] | 6.11 [5.58 to 6.68] | 2.39 [2.14 to 2.67]
Statistical Analysis 1: Comparison: THS 2.2 Menthol (mTHS 2.2) vs Menthol Conventional Cigarette (mCC); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on COHb levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 38.14, 95% CI 2-sided [34.24 to 42.47] — Geometric LS mean ratio mTHS 2.2:mCC

ADVERSE EVENTS:
Time Frame: From the informed consent form (ICF) signature until the end of the safety follow-up period, up to 150 days (including a screening period of up to 28 days, an 8-day confinement period followed by an 85-day ambulatory setting, and by a 28-day safety follow-up period (28 days after discharge of the subject or early discontinuation)).
Description: The adverse events and serious adverse events reported are for the post-randomization period.
  The safety was assessed in the safety population, consisting of 165 subjects: 160 randomized subjects (80 in mTHS 2.2, 41 in mCC and 39 in SA) and 5 subjects exposed to mTHS 2.2 from the product trial on Day -2 but not randomized. After randomization, the Safety Population consisted of 160 subjects with one valid post-randomization safety assessment.
Arm/Group | THS 2.2 Menthol (mTHS 2.2) | Menthol Conventional Cigarette (mCC) | Smoking Abstinence (SA)
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 31/80 | 12/41 | 16/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THS 2.2 Menthol (mTHS 2.2) (N=80) | Menthol Conventional Cigarette (mCC) (N=41) | Smoking Abstinence (SA) (N=39)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Blood triglycerides increased (Investigations) | 2 (2) | 2 (3) | 2 (2)
Haemoglobin decreased (Investigations) | 11 (14) | 4 (5) | 6 (8)
Lymphocyte count increased (Investigations) | 6 (7) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 3 (4)
Neutrophil count decreased (Investigations) | 4 (5) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Analysis of Primary Outcomes required data from the PP set at Baseline, Day 5 (MHBMA, 3-HPMA, S-PMA, and COHb), and Day 90 (Total NNAL). Differences in the number of participants for each outcome is due to missing data at baseline or at Day5/90.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specifies that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2014-04-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT01989156/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT01989156/SAP_001.pdf